CLINICAL TRIAL: NCT01270568
Title: Mind-body Interventions in Cardiac Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Jeff C. Huffman, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009P002386
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Acute Coronary Syndrome; Congestive Heart Failure
Keywords: positive psychology; cardiovascular disease
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure; Cardiovascular Diseases | interventions — Psychology, Positive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Positive Psychology (Experimental): 8 weekly positive psychology exercises
  Interventions: Other: Positive Psychology
- Relaxation Response (Active Comparator): Meditation-based treatment
  Interventions: Behavioral: Relaxation Response
- Recollection (Sham Comparator): Recollection of daily events, recorded weekly
  Interventions: Behavioral: Recollection

INTERVENTIONS:
Other: Positive Psychology — Weekly exercises focused on optimism, gratitude, altruism, and other positive affective states
  Arms: Positive Psychology
Behavioral: Relaxation Response — Daily practice of relaxation response, reviewed on a weekly basis
  Arms: Relaxation Response
Behavioral: Recollection — Subjects record daily events on a weekly basis for 8 weeks
  Arms: Recollection

SUMMARY:
This study is investigating whether a series of psychological exercises, called positive psychology, provides benefit to patients who have been hospitalized for heart disease (an 'acute coronary syndrome' or heart failure).

In this study, subjects are randomly assigned to complete 8 positive psychology exercises over 8 weeks, or to complete different exercises in control groups.

We hypothesize that patients who are assigned to the positive psychology tasks will be able to complete the exercises at a high rate, will feel that the exercises were easy to perform, and will have greater improvements of optimism, anxiety, mood, and health-related quality of life than subjects in the control conditions.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization at Massachusetts General Hospital for an acute coronary syndrome or congestive heart failure
* Able to read/write in English
* Have working home or cellular phone

Exclusion Criteria:

* Cognitive disorder
* Medical condition likely to lead to death within 6 months
* Illness leading to inabilty to consent or complete study exercises
* Current or prior participation in positive psychology interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Feasiblity | 8 weeks
  Percentage of exercises completed in the 8 week period

SECONDARY OUTCOMES:
Optimism | 8 weeks
  Self-report (on Likert scale) of optimism
Happiness | 8 week
  Score on Subjective Happiness Scale Score on Happiness subscale of CES-D
Depression | 8 weeks
  Center for Epidemiologic Studies Depression Scale (CES-D)
Anxiety | 8 weeks
  Hospital Anxiety and Depression Scale--Anxiety subscale
Mental-health related quality of life | 8 weeks
  SF-12 Mental Component Score

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States